CLINICAL TRIAL: NCT05571995
Title: Theory-Based Intervention Module on Occupational Safety and Health (TRIMOSH) in Improving Knowledge, Attitude, and Practice Among Food Industries Workers: Study Protocol for A Randomized Controlled Trial
Brief Title: RCT of TRIMOSH Module in Improving Knowledge, Attitude, and Practice Among Food Industries Workers
Acronym: TRIMOSH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Rahmat bin Dapari, Dr, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TRIMOSH
Record Dates: First submitted 2022-09-29; First posted 2022-10-07 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Occupational Injuries; Occupational Diseases
MeSH Terms: conditions — Occupational Injuries; Occupational Diseases | interventions — Health

STUDY DESIGN:
Intervention Model Description: single blinded cluster randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive TRIMOSH
  Interventions: Behavioral: TRIMOSH
- Control (No Intervention): The control group will receive no intervention.

INTERVENTIONS:
Behavioral: TRIMOSH — TRIMOSH will improve the knowledge, attitude and practice on occupational and health
  Other Names: Theory-Based Intervention Module on Occupational Safety and Health
  Arms: Intervention

SUMMARY:
Introduction: The food and beverages industry contributed a significant income to Malaysia's Gross Domestic Products. The contribution is projected to swell more in the upcoming years. As the industry expands, the demand for the workforce in the food premises will also continuously increase. They are exposed to risks arising from physical, chemical, biological, mechanical, and social hazards while performing their duties. Thus, it is essential for Food Industries Workers to be equipped with the proper knowledge, attitude, and practice (KAP) towards safety and health.

Methods and analysis: Theory Based Intervention Module on Occupational Safety and Health (TRIMOSH) is a single blinded, cluster randomized controlled trial study will be implemented among Food Industries Workers in Selangor, Malaysia. Partnering with the Food Handler Training School in Selangor, 10 pairs of Food Handler Training School with 12 participants per group (n = 240) will be recruited for balanced randomization intervention and control conditions. Data collection of all participants will be at enrollment, one months and three months. Generalized Linear Mixed Model (GLMM) will be conducted to determine the effects of intervention within and between study groups. Primary outcomes are to increase knowledge, attitude, and practice (KAP) and secondary outcome is safe practice score at food premise.

Ethic and Dissemination: his study has been submitted for approval by the Ethics Committee for Research involving Human Subject of Universiti Putra Malaysia (JKEUPM-2022-346). All participants will provide consent prior to participation. The results will be reported in international peer- reviewed journals and presented at conferences and other platforms.

DETAILED DESCRIPTION:
Food Industries workers are defined as individuals who are directly involved in the food preparation, come into contact with food or food contact surfaces, and handle packaged or unpackaged food, or appliances, on any food premises (1). Since 1996, the Ministry of Health Malaysia (MOH) has launched the food handler training course to give exposure and awareness to food Industries workers on food safety, hygiene, self-hygiene, and premise hygiene, mainly to prevent food poisoning incidents in the country (2). Subsequently, under Food Hygiene Regulations 2009, all food Industries workers are compulsory to attend the Food Handler Training Programme organized by any school or institute that has been certified by MOH. Under this regulation, any food industries workers who fails to undergo training or obtain a Certificate of Food Handlers Training shall be liable to a fine or compound not exceeding RM10,000 or imprisonment for a term not exceeding 2 years (3).

Regarding occupational safety and health of workers who work as food industries workers in Malaysia, they are generally governed and regulated by Act 514 Occupational Safety and Health (OSHA) Act 1994 as for any other occupations (4). It is within the spirit of the act to secure the safety, health, and welfare of persons at work to protect the workers and others from any risk or health implication associated with the activities of persons at work and prevent occupational diseases. An occupational disease is defined as any disease contracted due to exposure to risk factors arising from work activity (5). However, there is currently no occupational safety and health training module, required or made compulsory by the government for food industries workers to equip them with appropriate knowledge, attitude, and practice on occupational safety and health to prevent injuries and illnesses related to their work.

The food and beverages industry contributed a significant income to Malaysia's Gross Domestic Products (6). The contribution is projected to swell more in the upcoming years. As the industry expands, the demand for the workforce in the food premises will also continuously increase. The workforce substantially involves workers from the food processing sector, food distribution sector, and food service sector in the food premises. They are exposed to risks arising from physical, chemical, biological, mechanical, and social hazards while performing their duties. As the workers' volume increases, the number of accidental injuries or occupational diseases related to the food and beverages industry is expected to increase as well. Thus, it is essential for food industries workers who work in food premises to be equipped with the proper knowledge, attitude, and practice (KAP) towards safety and health.

At global level, 14.1% of nonfatal occupational injuries and illnesses involving days away from work (DAFW) in private Industry in 2020 goes to manufacturing industry including the food and beverages sector while 7.2% from food services (7).The highest number of nonfatal occupational injuries and illnesses involving days away from work (DAFW) in private Industry involving food industries workers within the industries contribute about 22% of total reported cases or around 0.3 million cases (8). Of all the reported injuries and illnesses cases, cuts, lacerations and punctures (15%) were the highest contributors of injuries and illnesses for known classified cases among food industries workers, followed by sprain, strains, and tears (15%), soreness and pain (13%), thermal burn (8%), bruises and contusions (5%), fractures (4%), multiple traumatic injuries (1%), chemical burns and corrosions (1%), carpal tunnel syndrome (1%), amputation (0.4%) and tendonitis (0.06%). However, there was a sum of reported cases that were non-classifiable and contributed to about 35% of the total reported cases among food industries workers (9). The highest number of injuries and illnesses experienced by food industries workers have resulted from exposure to harmful substances or environments (34%), followed by contact with objects or equipment (22%), falls, slips, and trips (21%), overexertion and bodily reaction (19%), transportation incidents (2%), violence and other injuries by persons or animal (1%), other events or exposures (0.4%) and fires and explosions (0.09%) (10). the top ten occupations that have been reported to have the highest incidence of occupational injuries and illnesses among food industries workers were observed among those who work in food preparation and serving related occupations (25%), cooks, and food preparation workers (10%), food and beverage serving workers (9%), food processing workers (6%), cooks (5%) fast food and counter workers (5%), food preparation workers (5%), supervisors of food preparation and serving workers (4%) butchers and other meat, poultry and fish processing workers (3%) and other food preparation and serving related workers (3%) (9).

Based on local statistics, the manufacturing industry, including the food and beverages sector, accounted for the most significant contributor to all confirmed occupational poisoning and disease cases at 82.3%. On the other hand, the percentage of confirmed cases from hotels and restaurants and wholesale and retail trades accounted for 0.5% and 0.3% of total confirmed cases. According to the sector, in terms of accidental injury at the workplace, DOSH Malaysia generally reported an increasing trend of accidents among food industries workers from year to year. In 2020 only, 62% of accidents with temporary disability, 84% of accidents with a permanent disability, and 34% of death reported to DOSH were coming from the manufacturing industry. On the other hand, 2% of accidents with temporary disability, 0.4% of accidents with a permanent disability, and 0.7% of death reported to DOSH came from the hotel and restaurants industry. Wholesale and retail trade reported a 2% of accidents with temporary disability, 0.4% of accidents with a permanent disability, and 0.4% of death to DOSH (5).

Although the Ministry of Health have introduced compulsory food h industries workers training course. This course was formalized and uniformed mainly on food aspect which is introduction, food hygiene, food safety, and critical factors of food poisoning. Based on the available data on occupational poisoning, occupational diseases, and accidents that lead to temporary and permanent disability among food industries workers, related training such as Theory-based Intervention Module on Occupational Safety and Health (TRIMOSH) is appropriate to be implemented for food industries workers to prevent such occurrences.

Study aims Our overarching objective is to create an effective safety and health program for Food Industries Workers to enhance their knowledge, attitude, and practice. The intervention was titled the TRIMOSH (Theory-Based Intervention Module on Occupational Safety and Health) Program. Investigators hypothesized that the intervention group would demonstrate beneficial effects related to the intended outcomes of safety and health (knowledge, attitude and practice score).

Methods Overview and timeline This research protocol details the process of development, implementation and effectiveness assessment of Theory-based Intervention Module on Occupational Safety and Health (TRIMOSH) among Food Industries Workers. The study will be conducted over 24 months, from October 2022 to October 2024. The study consists of two main phases, which are Phase I: Intervention module development, and Phase II: Implementation and effectiveness assessment of intervention module.

Phase I: Intervention module development A systematic step-by-step procedure will be conducted for designing Theory-based Intervention Module on Occupational Safety and Health (TRIMOSH). The intervention development will consist of seven steps as outlined below. To ensure that the objectives of TRIMOSH and Food Handlers Training Course is non overlapping, the participant and subject matter expert during TRIMOSH development will be emphasize that TRIMOSH will focus on Food Industries Workers safety and health while the usual Food Handler Training Course focus on food safety.

Step

1. Identification of safety and health problems, and intervention need
2. Priorities the safety and health problems
3. Develop prototype module focusing on the solution and target group
4. Decide the appropriate method and media for intervention
5. Pilot testing
6. Module evaluation
7. curriculum refinement

Phase II: Implementation and effectiveness assessment The TRIMOSH trial is a two-arm cluster randomised, single blinded, controlled, parallel trial. Partnering with the Food Handler Training School in Selangor, ten pairs of Food Handler Training School will be recruited for balanced randomization of groups to intervention and control conditions. One cluster define as one comparable Food Handler Training School. Intervention and control group will be assigned using a coin toss randomization technique. Cluster randomisation will be use in this study to avoid contamination between intervention and control group. The intervention group will receive TRIMOSH after completed food handler training course while the control group will receive the food handler training course as the usual current practice. The inclusion criteria for the participants will be Food Industries Workers registered under food handler training course, and never attend any occupational safety and health course. The exclusion criteria will be not able to read in local language (Bahasa Melayu) and non-Malaysian resident.

To increase the acceptance of the Food Industries Workers as well as stakeholder on this TRIMOSH, the duration and method of delivery will be identical with Food Handler Training Course which is four hours face to face training course.

Sample size A prior power analyses specified an enrolment target of 20 groups of 6 participants per condition. The average attrition rate across prior intervention studies was 20%, conservatively estimated attrition at 20% for each testing time point when designing the target sample size. The required sample size is 20 groups of 12 participants per group (N = 240). To motivate retention, the investogators plan lottery style drawings for participants who complete each date collection phase. the investigators also will provide retention bonus pay for those completed all four data collection phases.

Data collection Data collection for both intervention and control participants will be collected prior to the intervention (T0), at the end of intervention (T1), one month (T2) and three months (T3) post intervention.

Data analysis Quantitative Data will be compiled and analyzed using the statistical Package for the Social Science (IBM SPSS, Version 26.0). Descriptive statistics using continuous data will be presented using mean (Standard Deviation, SD) if normally distributed and median (interquartile range, IQR) if data not normally distributed. Categorical data will be presented in frequency and percentage.

Normality of data will be checked prior the analysis graphically and statistically. If the criteria for normally distributed data have been fulfilled, parametric tests will be used for further analysis, while non-parametric test will be used if the data not normally distributed. Missing value and irrelevant answers will be handled.

Generalized Linear Mixed Model (GLMM) will be conducted to determine the effects of sociodemographic factors (age, gender, ethnicity, level of education), socioeconomic (employment status, household income), working experience (duration) and previous training (training attended) on KAP on occupational safety and health at food premises among Food Industries Workers pre and post intervention within and between study groups.

The study protocol and all its procedures have been approved by the Ethics Committee for Research involving Human Subject of Universiti Putra Malaysia (JKEUPM-2022-346). All participants will be informed that their enrollment will in no way affect their relationship with their employer. Consent from each participant will be obtained using consent form upon agreement to participate in the study before answering the baseline questionnaire. Participants are allowed to withdraw at any point during the study.

Dissemination Research dissemination and knowledge translation will be conducted in three ways. First, the investigators will build on networking among stakeholder at national level to broader health policy in order to shape policy and improve the safety and health of food industries workers for wider dissemination nationally. Second, the investigators will engage with the Medical Doctor (MD), Occupational Health Doctor (OHD) and Safety and Health Officer (SHO) to inform them the progress and emerging research findings. Subsequently Train the Trainers (TTT) will be conducted among them to expand the TRIMOSH nationwide. Third, the investigators will also disseminate findings via traditional academic routes of conferences and peer-reviewed publications.

Consent for publication Consent from the participants for publication will be obtained from the same consent for participation. The full study publication approval will be obtained from the Director General of Ministry of Health Malaysia as part of the requirement as the participants come from food handler training course Ministry of Health.

ELIGIBILITY:
Inclusion Criteria:

* food industries workers registered under food handler training course,
* age 18-65 years

Exclusion Criteria:

* not able to read in local language (Bahasa Melayu)
* non-Malaysian resident.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
knowledge on occupational safety and health | 3 months
  Adopted, modified and validated knowledge score questionnaire on occupational safety and health will be used to meassure the knowledge level
attitude on occupational safety and health | 3 months
  Adopted, modified and validated attitude score questionnaire on occupational safety and health will be used to meassure the attitude level
practice on occupational safety and health | 3 months
  Adopted, modified and validated practice score questionnaire on occupational safety and health will be used to meassure the practice level

CONTACTS AND LOCATIONS:
Overall Officials: Rahmat Dapari, DrPH, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Universiti Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
We are committed to sharing the individual participant data (IPD) collected during the course of this study upon request, to promote transparency and scientific collaboration
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After 1st publication of completed study

REFERENCES:
- [Derived] Dapari R, Mahfot MH, Ahmad Zamzuri M'I, Md Isa Z, Hassan MR, Che Dom N, Syed Abdul Rahim SS. Theory-Based Intervention Module on Occupational Safety and Health (TRIMOSH) in improving knowledge, attitude, and practice among food industry workers: Study protocol for a randomised controlled trial. PLoS One. 2024 Jan 2;19(1):e0295771. doi: 10.1371/journal.pone.0295771. eCollection 2024. PMID 38165964